CLINICAL TRIAL: NCT04956900
Title: An Open Label, Multiple Ascending Dose Study of the Safety, Tolerability and Bio-effect of Aurase for Wound Debridement in Patients With Venous Leg Ulcers.
Brief Title: Clinical Trial Enzyme Application Targeting Venous Leg Ulcers
Acronym: CLEANVLU
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SolasCure Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SC-VLU-001; 2020-001392-32 (EudraCT Number)
Record Dates: First submitted 2021-06-25; First posted 2021-07-09 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Venous Leg Ulcer; Leg Injuries and Disorders
Keywords: Wounds; Chronic Leg Ulcer; Leg Ulcer; Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer; Leg Injuries; Disease; Wounds and Injuries; Leg Ulcer

STUDY DESIGN:
Intervention Model Description: Cohort study design with each cohort having an ascending dose of Aurase wound gel. At the time of initiation, 5 sequential cohorts are planned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Aurase wound gel X0 (Experimental): Cohort 1: Aurase wound gel x0 dose concentration
  Interventions: Drug: Aurase Wound gel
- Aurase wound gel X1 (Experimental): Cohort 2: Aurase wound gel x1 dose concentration
  Interventions: Drug: Aurase Wound gel
- Aurase wound gel X1.8 (Experimental): Cohort 3: Aurase wound gel X1.8 dose concentration
  Interventions: Drug: Aurase Wound gel
- Aurase wound gel X5 (Experimental): Cohort 4: Aurase wound gel X5 dose concentration
  Interventions: Drug: Aurase Wound gel
- Aurase wound gel X9 (Experimental): Cohort 5: Aurase wound gel X9 dose concentration
  Interventions: Drug: Aurase Wound gel

INTERVENTIONS:
Drug: Aurase Wound gel — Aurase Wound Gel is reconstituted from Aurase Component A (a hydrogel) and Aurase Component B (stabilised solutions of Aurase enzyme). By diluting different strengths of Aurase Component B with Component A, specific concentrations of Aurase Wound Gels with differing Aurase contents are yielded.

SUMMARY:
This is an adaptive open-label, first-in-human (Phase IIa) study designed to assess the safety (and efficacy) of Aurase Wound Gel, an enzymatic debridement product, intended for topical application to sloughy venous leg ulcers (VLU)

DETAILED DESCRIPTION:
The study has been designed as a dose escalation study, and will serially explore increasing concentrations of the Aurase enzyme in a relevant patient population. Five cohorts (of 10 patients each, except cohort 1 with 5 patients), will receive standard of care supplemented with increasing concentrations of Aurase and will be assessed for clinical tolerability at the wound site, systemic safety and efficacy (extent of wound debridement) over a period of 4 weeks. Patients will receive a total of 12 doses of Aurase Wound Gel. At the end of the study, patients will revert to standard of care only.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18 years and older at screening
* Patients with at least one defined Venous Leg Ulcer (VLU) suitable for treatment that is no smaller than 2cm2 but no larger than 50cm2
* Presence of devitalised tissue within the reference ulcer suitable for debridement therapy
* Confirmed, clinically diagnosed VLU (30 days or more) which has been present for less than 2 years
* Willing and able to attend and comply with study visits and study related activities

Exclusion Criteria:

* Diabetic Foot Ulcer
* A clinical history of a bleeding disorder including haemophilia, purpura, or thrombocytopenia
* Current or history of use of anti-thrombotic therapy less than 7 days prior to screening.
* Stage 4 or 5 chronic kidney disease, defined as estimated glomerular filtration rate (eGFR) less than or equal to 30 mL/min
* Reference ulcer has active infection or florid oedema at screening
* Oral or intravenous antibiotics for any indication within 72 hours of screening
* Reference ulcer has exposed tendons, ligaments, muscle, or bone
* Active osteomyelitis, cellulitis or gangrene in either leg
* Patients with amputation above a trans metatarsal amputation (TMA) in the target leg
* Planned vascular surgery, angioplasty, or thrombolysis procedures within the study period, or 4 weeks before screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | From the time of signing informed consent up to the last visit (Day 29)
Change in study wound pain burden from baseline measured by Numerical Rating Scale (NRS) | Pre-dosing and post-dose at day 1 (baseline) through to day 29 (end of study)
  Subject will be asked to describe the level of wound pain on a scale of 0-10: 0 being no pain, 10 being worst imaginable pain
Change in study wound itch burden from baseline measured by Numerical Rating Scale (NRS) | Pre-dose at day 1 (baseline) through to day 29 (end of study)
  Subject will be asked to describe the level of wound itch on a scale of 0-10: 0 being no itch, 10 being worst imaginable itch
Grading of clinical signs of wound inflammation | Pre-dosing and Post-dose at day 1 (baseline) through to day 29 (end of study)
  5-point ordinal grading scale (1 [none] to 5 [severe] ) of wound erythema, oedema made by clinical assessor by Visual Assessment (VA)
Grading of clinical signs of wound infection | Day 1 (baseline) through to day 29 (end of study)
  5-point ordinal grading scale (1 [none] to 5 [severe] ) of wound exudate and induration or grading of presence/absence of wound bleeding and infection made by clinical assessor by Visual Assessment (VA)

SECONDARY OUTCOMES:
Change in surface area of wound compared to baseline | Day 1 (baseline), day 5, day 12, day 19, day 29 (end of study)
Change in surface area of devitalised tissue (slough, eschar) compared to baseline | Day 1 (baseline), day 5, day 12, day 19, day 29 (end of study)
Change in surface area of granulation tissue from baseline | Day 1 (baseline) , day 5, day 12, day 19, day 29 (end of study)
Number of patients achieving 100% debridement | Day 1 (baseline), day 5, day 12, day 19, day 29 (end of study)
  Determination of 100% debridement made by clinical assessor upon assessment of wound at each study visit
Systemic absorption of Aurase enzyme assessed through pharmacokinetic profiling of blood samples | Pre-dose and Post dose at day 1 (baseline) and day 29 (end of study) or early termination visit (if applicable)
Assessment of the presence of antibodies to Aurase in plasma (Anti-Drug Antibody [ADA] activity) through applicable laboratory analysis of blood samples | Day 1 (Baseline) and day 29 (end of study) or early termination visit (if applicable)
Assessment of systemic clotting factors in plasma | Day 0 (Screening), day 1 (Baseline), day 8 and day 29 (end of study) or early termination visit (if applicable)
  Activated partial thromboplastin time (APTT)/ prothrombin time (PT)/Fibrinogen plasma concentrations determined through laboratory analysis of blood samples

CONTACTS AND LOCATIONS:
Locations (8):
- United States (5):
  - Center for Clinical Research, San Francisco, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Doctors Research Network, Miami, Florida
  - University of Miami, Miami, Florida
  - FASMA, Salem, Virginia
- Hungary (2):
  - Óbudai Egészségügyi Centrum Kft., Budapest
  - Uno Medical Trials, Budapest
- Hull Royal Infirmary, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: No